CLINICAL TRIAL: NCT02859207
Title: An Open-Label Parallel-Group Study to Evaluate the Pharmacokinetics of E2609 and Its Metabolites in Subjects With Mild and Moderate Hepatic Impairment Compared With Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of E2609 and Its Metabolites in Subjects With Mild and Moderate Hepatic Impairment Compared With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2609-A001-103
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Early Alzheimer's Disease
Keywords: Early Alzheimer's disease; E2609; Mild and Moderate Hepatic Impairment
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Participants with mild hepatic impairment (Child-Pugh class A).
  Interventions: Drug: E2609
- Cohort 1C (Experimental): Healthy participants (control) matched to participants in Cohort 1.
  Interventions: Drug: E2609
- Cohort 2 (Experimental): Participants with moderate hepatic impairment (Child-Pugh class B)
  Interventions: Drug: E2609
- Cohort 2C (Experimental): Healthy participants (control) matched to participants in Cohort 2
  Interventions: Drug: E2609

INTERVENTIONS:
Drug: E2609 — Participants will receive a single 50-mg dose (1× 50-mg E2609 tablet).

SUMMARY:
The primary objective of the study is to evaluate the effects of hepatic impairment on the pharmacokinetics (PK) of E2609 after a single dose administration.

ELIGIBILITY:
Inclusion Criteria

1. Nonsmoking, male or female, ≥18 years and ≤70 years of age at the time of informed consent, and with body mass index (BMI) of up to 40 kg/m2, inclusive.
2. For Cohorts 1 and 2: stable mild or moderate hepatic impairment conforming to Child-Pugh class A or B, respectively, documented by medical history, physical examination and 1 or more of the following diagnostic procedures documented in the medical notes: liver biopsy, computed tomography (CT) scan, magnetic resonance imaging (MRI), ultrasound, radionuclide liver/spleen scan, or abdominal laparoscopy. Participants whose liver imaging was done more than 1 year ago or previous results were not available, should have a liver ultrasound scan to ensure that the liver structure is consistent with the diagnosis of hepatic impairment and that there are no exclusionary features.
3. For Cohorts 1C and 2C: healthy participants matched to participants with mild or moderate hepatic impairment with regard to age (±10 years), body weight (±20%), and gender; and as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECG), and clinical laboratory determinations.

Exclusion Criteria

For all Participants (Cohorts 1, 2, 1C, and 2C)

1. Females participants who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] test. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the dose of study drug.
2. Females of childbearing potential who:

   * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation.
   * Are currently abstinent and do not agree to use a double-barrier method (as previously described) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation .
   * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product except those containing estradiol for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation.
   * Are using estradiol-containing hormonal contraceptives within 4 weeks before dosing (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [eg, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy; all with surgery at least 1 month before dosing]).
3. Males who have not had a successful vasectomy (unconfirmed azoospermia) or they and their female partners do not meet the criteria specified in exclusion criterion 2 (eg, unwilling to refrain from sexual activity, not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation).
4. Inability to tolerate oral medication.
5. Inability to be venipunctured and/or tolerate venous access. For Hepatically Impaired Participants (Cohorts 1 and 2)
6. Any significant acute medical illness (such as new conditions or exacerbation or pre-existing conditions) within 4 weeks before dosing.
7. Medical conditions which are not adequately and stably controlled on stable doses of medications or which, in the clinical opinion of the investigator, may interfere with study procedures or participant safety within 4 weeks before dosing; eg, psychiatric disorders and disorders of the gastrointestinal tract, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism. Participants with history of seizures during adulthood are excluded. Participants with a history of Gilbert's syndrome are excluded.
8. History of esophageal and gastric variceal bleeding within the past 3 months unless the participant has completed a course of endoscopic therapy with the appropriate documentation (eg, endoscopy report) of successful ablation of esophageal varices; participants with esophageal varices may be included if not bleeding within the past 3 months or have been treated adequately by ablation therapy.
9. Spontaneous bacterial peritonitis within 3 months before dosing.
10. Treatment with plasmapheresis within 6 months before dosing.
11. Primarily cholestatic liver diseases (eg, primary biliary cirrhosis or primary sclerosing cholangitis).
12. Current or recent (within 3 months before Screening) history of significant gastrointestinal disease other than that secondary to hepatic impairment.
13. Autoimmune liver disease.
14. Active alcoholic hepatitis determined either clinically or by histology per the discretion of the investigator.
15. History of hepatoma or metastatic disease of the liver.
16. Presence of severe ascites or edema.
17. Presence of hepatopulmonary syndrome or hydrothorax, or hepatorenal syndrome.
18. Known significant bleeding diathesis that could preclude multiple venipunctures (International Normalized Ratio [INR] >2.5).
19. Any major surgery within 4 weeks before dosing.
20. Any history of abdominal surgery that may affect the pharmacokinetic (PK) of E2609 (eg, hepatectomy, nephrectomy, digestive organ resection, transjugular intrahepatic portosystemic shunt [TIPS]) at Screening or Baseline (history of cholecystectomy need not be exclusionary).
21. Donation of blood or plasma within 4 weeks before dosing.
22. Receipt of blood or blood products within 4 weeks before dosing.
23. Known to be human immunodeficiency virus (HIV)-positive at Screening.
24. Creatinine clearance <60 mL/min at Screening or Baseline, as calculated using Cockroft and Gault equation.
25. Known history of clinically significant drug allergy at Screening.
26. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening.
27. History of drug or alcohol dependency or abuse within 4 weeks before Screening, or those who have a positive urine drug test or breath (or urine) alcohol test at Screening or Baseline unless a prescribed medication for the underlying condition is the cause of the positive urine screen.
28. A prolonged QT/QTc interval (QTc Fridericia [QTcF] >480 ms) demonstrated on the ECG at Screening or Baseline. A history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome).
29. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5× the half-life of the investigational drug, whichever is longer, preceding informed consent.
30. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], and charbroiled meats) within 1 week before dosing.
31. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing .
32. Engagement in strenuous exercise within 2 weeks before Baseline.

    For Healthy Participants (Cohorts 1C and 2C)
33. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
34. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system), or participants who have a congenital abnormality in metabolism. Participants with history of seizures in adulthood are excluded.
35. Any history of gastrointestinal surgery that may affect the drug absorption (eg, hepatectomy, nephrotomy, digestive organ resection, but not cholecystectomy) at Screening.
36. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital sign assessments, ECG finding, or laboratory test results that require medical treatment at Screening.
37. A prolonged QT/QTc interval (QTcF >450 ms) demonstrated on ECG at Screening or Baseline. A history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome), or the use of concomitant medications that prolonged the QT/QTc interval.
38. Known history of clinically significant drug allergy at Screening.
39. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening.
40. Known to be HIV-positive at Screening.
41. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening.
42. History of drug or alcohol dependency or abuse within the 1 year before Screening, or those who have a positive urine drug test or breath (or urine) alcohol test at Screening or Baseline.
43. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], and charbroiled meats) within 1 week before dosing.
44. Intake of herbal preparations containing St. John's wort within 4 weeks before dosing.
45. Use of prescription drugs except those allowed per the inclusion/exclusion criteria (eg, contraception) within 4 weeks or 5 half-lives, whichever is longer, before dosing.
46. Intake of over-the-counter (OTC) medications within 2 weeks or 5 half-lives, whichever is longer, before dosing.
47. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5x the half-life of the investigational drug, whichever is longer, preceding informed consent.
48. Receipt of blood or blood products within 4 weeks, or donation of blood within 4 weeks, of dosing.
49. Engagement in strenuous exercise within 2 weeks before Baseline.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Mean maximum plasma concentration (Cmax) of E2609 | Day 1 through 7
  Blood samples for pharmacokinetic (PK) assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean area under plasma concentration versus time curve from time zero to time of last quantifiable concentration (AUC(0-t)) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean area under plasma concentration versus time curve from time zero to infinity (AUC(0-inf)) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).

SECONDARY OUTCOMES:
Mean time to reach maximum plasma concentration (tmax) of E2609 and its metabolites | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean terminal phase plasma half-life (t1/2) of E2609 and its metabolites | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean apparent total body clearance (CL/F) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean apparent volume of distribution (Vz/F) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean ratio of AUC(0-inf) of individual metabolite to AUC(0-inf) of E2609, corrected for molecular weight (AUC metabolite ratio) | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean plasma protein unbound fraction (fu) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean Cmax values adjusted for unbound fraction in plasma (Cmaxu) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean AUC(0-inf) values adjusted by unbound fraction in plasma (AUCu) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Mean Apparent clearance relative to the unbound plasma concentration based on AUCu (CLu/F) of E2609 | Day 1 through 7
  Blood samples for PK assessments will be collected on Day 1 (before dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after dosing), Day 2 (24 and 36 hours after dosing), Day 3 (48 hours after dosing), Day 4 (72 hours after dosing), Day 5 (96 hours after dosing), Day 6 (120 hours after dosing), and Day 7 (144 hours after dosing).
Number of participants with treatment emergent adverse events and serious adverse events | Up to approximately 36 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota